CLINICAL TRIAL: NCT01021865
Title: Effects of Hyperglycemia on Myocardial Perfusion in Humans With and Without Type 2 Diabetes: Modulation by Glucagon-Like-Peptide-1
Brief Title: Effects of Hyperglycemia on Myocardial Perfusion in Humans With and Without Type 2 Diabetes
Acronym: GLP-1
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: University of Nebraska (Other); Astellas Pharma US, Inc. (Industry); Lantheus Medical Imaging (Industry)
Responsible Party: Principal Investigator, Sharon Mulvagh, PI, Mayo Clinic
Other Study IDs: 08-008750
Record Dates: First submitted 2009-10-30; First posted 2009-11-30 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus Type 2
Keywords: GLP-1; Myocardial contrast echocardiography; Myocardial perfusion
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2 | interventions — regadenoson; perflutren

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- With type 2 Diabetes
  Interventions: Drug: Glucagon-Like-Peptide-1/Regadenoson/Perflutren Lipid Microsphere
- Without type 2 diabetes
  Interventions: Drug: Glucagon-Like-Peptide-1/Regadenoson/Perflutren Lipid Microsphere

INTERVENTIONS:
Drug: Glucagon-Like-Peptide-1/Regadenoson/Perflutren Lipid Microsphere — GLP-1 at a rate of 1.2 pmol/kg/min
  Regadenoson as a stress agent 0.4mg IV given during MCE
  Definity:0.6 ml of Definity diluted with 30ml of 0.9% saline infused by SYRINGE Infusion Pump
  Other Names: Lexiscan; Definity

SUMMARY:
The overall goal of this proposal is to determine the effects of acute hyperglycemia and its modulation by Glucagon-like Peptide-1 (GLP-1) on myocardial perfusion in type 2 diabetes (DM). This study plan utilizes myocardial contrast echocardiography (MCE) to explore a) the effects of acute hyperglycemia on myocardial perfusion and coronary flow reserve in individuals with and without DM; and b) the effects of GLP-1 on myocardial perfusion and coronary flow reserve during euglycemia and hyperglycemia in DM. The investigators will recruit individuals with and without DM matched for age, gender and degree of obesity. The investigators will measure myocardial perfusion at rest and during vasodilator stress (to ascertain coronary flow reserve) while subjects are under controlled pancreatic clamp conditions during euglycemia (glucose ~100 mg/dl) and hyperglycemia (glucose ~250 mg/dl) in the presence and absence of concomitant GLP-1 infusion. The investigators believe that the translational significance of their studies is immense, impacting upon both acute and chronic cardiovascular disease manifestations. The effect of glycemic control on cardiovascular outcomes, morbidity and mortality remains an area of active investigation, fueled by the recent conflicting results of several large clinical trials (ACCORD, United Kingdom Prospective Diabetes Study (UKPDS), ADVANCE, VADT). If the investigators find that hyperglycemia is associated with altered myocardial perfusion, the mechanistic implications in the prevention and management of acute and chronic cardiovascular diseases in DM will be groundbreaking. Furthermore, if GLP-1 augments myocardial perfusion (as it does in the peripheral vasculature), the therapeutic benefits for prevention of cardiovascular events in this predisposed population are clear.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 40-60 years
* BMI< or = 35 kg/m2
* Diabetic subjects with HbA1c concentrations of < or = 8%.
* Diabetic subjects will be either on diet and lifestyle therapy alone, or monotherapy with metformin or sulphonylureas (except glyburide).
* All diabetic subjects should be on stable dose oral agent therapy for 3 months prior to enrollment.

Exclusion Criteria:

* Subjects with cerebrovascular or peripheral vascular disease.
* Subjects with suspected or overt autonomic neuropathy.
* Diabetic subject on thiazolidinediones, insulin, GLP-1 based therapies (exenatide or sitagliptin), alpha-glucosidase inhibitors, glyburide or combination antidiabetic drug therapies.
* Diabetics with microalbuminuria.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 25 subjects with type 2 diabetes and 25non-diabetic subjects matched for age, gender and degree of obesity will be studied.
  The diabetic subjects will be between 40 and 60 years of age and will have a body mass index of < or =35 kg/m2. Diabetic subjects treated according to ADA guidelines will be eligible for study including a blood pressure < 140/90, LDL cholesterol < 130 mg/dl, HDL cholesterol >40 mg/dl and triglycerides <200 mg/dl.
  All nondiabetic subjects will not have a history of diabetes in their first degree family members. None of the subjects will have any overt evidence of cardiac, renal, pulmonary or hepatic disorder nor will they be engaging in regular vigorous physical activities. All subjects will undergo a resting ECG and a treadmill ECG test to ensure that they do not have active or occult coronary artery disease unless such testing had been completed within six months of enrollment and reported as normal.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2010-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To determine whether hyperglycemia alters myocardial perfusion in subjects with type 2 diabetes | Nov 2009-2011

SECONDARY OUTCOMES:
To determine whether GLP-1 modulates myocardial perfusion in subjects with type 2 diabetes. | Nov 2009-2011

CONTACTS AND LOCATIONS:
Overall Officials: Ananda Basu, MBBS, M.D., Principal Investigator — Mayo Clinic; Sharon L Mulvagh, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Abdelmoneim SS, Hagen ME, Mendrick E, Pattan V, Wong B, Norby B, Roberson T, Szydel T, Basu R, Basu A, Mulvagh SL. Acute hyperglycemia reduces myocardial blood flow reserve and the magnitude of reduction is associated with insulin resistance: a study in nondiabetic humans using contrast echocardiography. Heart Vessels. 2013 Nov;28(6):757-68. doi: 10.1007/s00380-012-0305-y. Epub 2012 Nov 23. PMID 23180239